CLINICAL TRIAL: NCT02022085
Title: Post-market Clinical Follow-up of a Magnetic Bone Conduction Implant (Cochlear Baha Attract System)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cochlear Bone Anchored Solutions (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CBAS5477
Record Dates: First submitted 2013-12-16; First posted 2013-12-27 (Estimated); Results first posted 2016-12-09 (Estimated); Last update posted 2018-10-12 (Actual); Status verified 2018-10

CONDITIONS: Deafness; Hearing Loss; Hearing Loss, Conductive
MeSH Terms: conditions — Deafness; Hearing Loss; Hearing Loss, Conductive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Baha Attract System (Experimental): This transcutaneous solution is based on a magnet coupling using magnets on both side of the skin;
  * One implant magnet
  * One external magnet on which a sound processor is attached, i.e. the Sound Processor magnet (SP magnet)
  Interventions: Device: Baha Attract System

INTERVENTIONS:
Device: Baha Attract System — The Cochlear Baha Attract System incorporates both implantable and external parts. The implantable parts include the BI300 Implant and the BIM400 Implant Magnet, which is intended to be fixated to the BI300 Implant. The external parts include the Sound Processor Magnet (SP Magnet), which, together with the Implant Magnet, constitute the transcutaneous coupling. The SP Magnet incorporates a soft material (Soft pad) at the tissue facing surface that is designed to distribute the pressure over the skin. The Baha Sound Processor attaches to the SP Magnet via a snap coupling.

SUMMARY:
The rationale behind this post-market clinical follow-up investigation is to collect data regarding the usability and clinical performance of the Baha Attract System in subjects with hearing impairment that are candidates for Baha surgery:

* to evaluate the efficacy of the Baha Attract System in terms of hearing performance compared to the unaided situation and compared to a pre-operative test situation using the sound processor on a Baha Softband;
* to evaluate the mid- and long-term safety of the Baha Attract System.

DETAILED DESCRIPTION:
This investigation was designed to collect data regarding the usability and clinical performance of the Baha Attract System in subjects with hearing impairment that were candidates for Baha surgery.

The investigation was performed in an open design since it was not possible to perform the investigation in a blinded fashion. The main evaluations of the investigation, i.e. free-field hearing tests, are standard audiological procedures that are routinely used in daily clinical practice at hospitals worldwide for evaluation of hearing performance in hearing impaired patients. The primary efficacy evaluation, audiometric thresholds, renders comparable results across different sites and countries as it is not a language-specific test. Language-specific audiological tests were performed as secondary efficacy evaluations; to enable comparison of data across sites, validated word lists were used at all sites and equivalent speaker configurations (speech from front, noise from behind) and test procedures (same noise and adaptive speech levels, etc) were used.

For the primary evaluation in the investigation, the Baha Attract System was compared to the pre-operative unaided situation, as the intended use of the system is to improve hearing performance in patients with conductive or mixed hearing loss or single-sided sensorineural deafness. Audiological test results with the Baha Attract System were also compared against results obtained with the same Sound Processor on a Baha Softband. Use of the Sound Processor on a Softband is a standard procedure that is routinely used as a pre-operative test prior to bone conduction hearing implant surgery. The Softband test allows the patient to pre-operatively experience hearing through the Sound Processor to get an indication of the post-operative hearing outcome and to choose a suitable Sound Processor.

The generic and hearing-specific quality of life questionnaires used in the investigation (HUI3, APHAB, SSQ) are validated scales that have been frequently used and reported in the literature.

ELIGIBILITY:
Inclusion Criteria:

Adult subject, i.e. ≥ 18 years of age

Conductive or mixed hearing loss in the ear to be implanted:

Bone conduction thresholds with a pure tone average PTA4 of < 30 dB hearing level (mean of 500, 1000, 2000 and 4000 Hz).

OR

Single-sided sensorineural deafness (SSD):

European sites: Bone conduction thresholds with a pure tone average PTA4 of < 30dB hearing level (mean of 500, 1000, 2000 and 4000 Hz) in the good ear.

US sites: Air conduction thresholds with a pure tone average PTA4 of 20 dB hearing level (mean of 500, 1000, 2000 and 3000 Hz) in the good ear OR Subject is indicated for an AC CROS but-for some reason-cannot or will not use an AC CROS.

No previous bone conduction implant on the side of the skull to be implanted. Signed informed consent.

Exclusion Criteria:

Subjects that are scheduled for simultaneous bilateral implant surgery. The investigation is limited to subjects with unilateral use of the Baha Attract System (however, bilateral hearing loss is not an exclusion criterion).

Suitable implant position for the BI300 Implant (4 mm or 3 mm) not found during surgery due to insufficient bone quality and/or bone thickness.

Less than 3 mm soft tissue thickness at the planned implant site. Subjects that have received radiation therapy at the same side of the skull where the Baha Attract System will be positioned.

Condition that could jeopardise osseointegration and/or wound healing as judged by the investigator (e.g. osteoporosis, psoriasis, use of corticosteroids).

Uncontrolled diabetes as judged by the investigator. Condition that may have an impact on the outcome of the investigation as judged by the investigator.

Unable to follow investigational procedures (e.g. to complete quality of life scales).

Participation in another investigation with pharmaceuticals and/or medical device.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2014-06; Primary Completion 2016-02 (Actual); Study Completion 2017-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Johan Blechert, M.Sc, Study Director — Cochlear Bone Anchored Solutions AB
Locations (6):
- United States (2):
  - Dr. Doug Backhus, Seattle, Washington
  - Christina Runge, Milwaukee, Wisconsin
- Dr. Myrthe Hol, Nijmegen, Netherlands
- World Hearing Center Institute of Physiology and Pathology of Hearing, Kajetany, Nadarzyn, Poland
- United Kingdom (2):
  - Peter Monksfield, Birmingham
  - Kevin Green, Manchester

RESULTS

PARTICIPANT FLOW:
Groups:
- Baha Attract System: This transcutaneous solution is based on a magnet coupling using magnets on both side of the skin;
  * One implant magnet
  * One external magnet on which a sound processor is attached, i.e. the Sound Processor magnet (SP magnet)
  Baha Attract System: The Cochlear Baha Attract System incorporates both implantable and external parts. The implantable parts include the BI300 Implant and the BIM400 Implant Magnet, which is intended to be fixated to the BI300 Implant. The external parts include the Sound Processor Magnet (SP Magnet), which, together with the Implant Magnet, constitute the transcutaneous coupling. The SP Magnet incorporates a soft material (Soft pad) at the tissue facing surface that is designed to distribute the pressure over the skin. The Baha Sound Processor attaches to the SP Magnet via a snap coupling.
Period: Overall Study
Arm/Group | Baha Attract System
Started | 54
Completed | 53
Not Completed | 1

BASELINE CHARACTERISTICS:
Population: ITT population, includes all subjects who received the surgical intervention.
Arm/Group | Baha Attract System
Number analyzed (Participants) | 54
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.1 (13.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 33
  Male | 21
Region of Enrollment [Number; unit: participants]
  Netherlands | 23
  United States | 1
  Poland | 14
  United Kingdom | 16
Type of hearing loss [Number; unit: participants]
  Conductive hearing loss | 39
  Single-sided sensorineural deafness | 15

OUTCOME MEASURES:

1. Primary Outcome: Hearing Performance: Threshold Audiometry PTA4: Unaided Versus Baha Attract
Description: The change of hearing performance with the Baha Attract System (aided) at 6, 12 and 24 months from the unaided hearing performance before surgery; measured as free-field hearing tests: Threshold audiometry PTA4 (mean of 500, 1000, 2000 and 4000 Hz).
  The units reported for PTA4 are decibels (dB). As such, a lower or more negative score is more desirable and reflects the ability to hear softer sounds.
Time Frame: Baseline (unaided) before surgery, 6, 12 and 24 months after surgery
Population: Intention-to-Treat (ITT) population; includes all subjects who received the surgical intervention.
Measure: Mean (Standard Deviation); unit: dB
Arm/Group | Baha Attract System
Number analyzed (Participants) | 54
dB
  PTA4 6 months, Baha Attract vs Unaided | -21.0 (10.4)
  PTA4 12 months, Baha Attract vs Baha Attract: number analyzed (Participants) | 52
  PTA4 12 months, Baha Attract vs Baha Attract | -20.9 (10.4)
  PTA4 24 months, Baha Attract vs Unaided: number analyzed (Participants) | 46
  PTA4 24 months, Baha Attract vs Unaided | -21.5 (8.3)
Statistical Analysis 1: Comparison: Baha Attract System; PTA4 6 months with Baha Attract vs Unaided; Test type: Superiority or Other; p < 0.0001, Fisher's non-parametric permutation test
Statistical Analysis 2: Comparison: Baha Attract System; PTA4 12 months with Baha Attract vs Unaided; Test type: Superiority or Other; p < 0.0001, Fisher's non-parametric permutation test
Statistical Analysis 3: Comparison: Baha Attract System; PTA4 24 months with Baha Attract vs Unaided; Test type: Superiority or Other; p < 0.0001, Fisher's non-parametric permutation test

2. Primary Outcome: Hearing Performance: Change in Threshold Audiometry: Unaided Versus Baha Attract
Description: The change of hearing performance with the Baha Attract System (aided) from the unaided hearing performance before surgery; measured as free-field hearing tests: Threshold audiometry PTA4 (mean of 500, 1000, 2000 and 4000 Hz).
  The units reported for PTA4 are decibels (dB). As such, a lower or more negative score is more desirable and reflects the ability to hear softer sounds.
Time Frame: Baseline (unaided) before surgery, 24 months after surgery
Population: Intention-to-Treat population (ITT); includes all subjects who received the surgical intervention.
Measure: Mean (Standard Deviation); unit: dB
Arm/Group | Baha Attract System
Number analyzed (Participants) | 46
dB
  Change of Threshold value at 250 Hz: number analyzed (Participants) | 45
  Change of Threshold value at 250 Hz | -19.9 (11.0)
  Change of Threshold value at 500 Hz | -25.3 (9.6)
  Change of Threshold value at 1000 Hz | -28.0 (12.4)
  Change of Threshold value at 2000 Hz | -19.6 (11.8)
  Change of Threshold value at 3000 Hz | -18.4 (10.9)
  Change of Threshold value at 4000 Hz | 13.2 (12.0)
  Change of Threshold value at 6000 Hz: number analyzed (Participants) | 45
  Change of Threshold value at 6000 Hz | -8.67 (8.88)
Statistical Analysis 1: Comparison: Baha Attract System; Baha Attract after 24 months vs Unaided situation Pre-Op; Test type: Superiority or Other; p < 0.0001, Fisher's non-parametric permutation test — All comparisons to the Unaided situation were p=<0.0001

3. Primary Outcome: Hearing Performance: Change in Threshold Audiometry: Unaided Versus Baha Attract
Description: The change of hearing performance with the Baha Attract System (aided) from the unaided hearing performance before surgery; measured as free-field hearing tests: Threshold audiometry at frequencies of 250, 500, 1000, 2000, 3000, 4000 and 6000 Hz).
  The units reported for threshold audiometry are decibels (dB). As such, a lower or more negative score is more desirable and reflects the ability to hear softer sounds.
Time Frame: Baseline (unaided) before surgery, 12 months after surgery
Population: Intention-to-Treat population (ITT); includes all subjects who received the surgical intervention.
Measure: Mean (Standard Deviation); unit: dB
Arm/Group | Baha Attract System
Number analyzed (Participants) | 51
dB
  Change of Threshold value at 250 Hz | -18.5 (14.3)
  Change of Threshold value at 500 Hz | -26.0 (13.0)
  Change of Threshold value at 1000 Hz | -26.5 (14.2)
  Change of Threshold value at 2000 Hz | -18.5 (13.5)
  Change of Threshold value at 3000 Hz | -16.3 (13.2)
  Change of Threshold value at 4000 Hz | -12.5 (12.2)
  Change of Threshold value at 6000 Hz | -7.25 (11.19)
Statistical Analysis 1: Comparison: Baha Attract System; Baha Attract after 12 months vs Unaided situation Pre-Op; Test type: Superiority or Other; p < 0.0001, Fisher's non-parametric permutation test — All comparisons to the Unaided situation were p=<0.0001

4. Primary Outcome: Hearing Performance: Change in Threshold Audiometry: Unaided Versus Baha Attract
Description: The change of hearing performance with the Baha Attract System (aided) from the unaided hearing performance before surgery; measured as free-field hearing tests:
  Threshold audiometry at individual frequencies 250, 500, 1000, 2000, 3000, 4000 and 6000 Hz.
  The units reported for threshold audiometry are decibels (dB). As such, a lower or more negative score is more desirable and reflects the ability to hear softer sounds.
Time Frame: Baseline (unaided) before surgery, 6 months after surgery
Population: Intention-to-Treat population (ITT); includes all subjects who received the surgical intervention.
Measure: Mean (Standard Deviation); unit: dB
Arm/Group | Baha Attract System
Number analyzed (Participants) | 54
dB
  Change of Threshold value at 250 Hz | -16.9 (12.9)
  Change of Threshold value at 500 Hz | -26.6 (12.8)
  Change of Threshold value at 1000 Hz | -26.4 (14.1)
  Change of Threshold value at 2000 Hz | -18.7 (12.1)
  Change of Threshold value at 3000 Hz | -16.9 (12.7)
  Change of Threshold value at 4000 Hz | -12.3 (10.6)
  Change of Threshold value at 6000 Hz | -7.04 (8.61)
Statistical Analysis 1: Comparison: Baha Attract System; Baha Attract after 6 months vs Unaided situation Pre-Op; Test type: Superiority or Other; p < 0.0001, Fisher's non-parametric permutation test — All comparisons to the Unaided situation were p=<0.0001

5. Secondary Outcome: Adaptive Speech Recognition in Noise Ratio: Unaided Versus Baha Attract
Description: The change of hearing performance with the Baha Attract System compared to the pre-operative unaided situation; Adaptive speech recognition in noise measured as signal to noise ratio
  The adaptive speech test in noise was conducted using validated lists of phonetically balanced sentences, with speech presented from the front (0 degrees azimuth) and noise from the back (180 degrees azimuth). The noise was kept constant at 65 dB SPL, and the speech was adapted in 2 dB steps to establish the speech-to-noise ratio (SNR) providing a 50% level of understanding.
  A ratio of 1 reflects the ability to correctly hear sentences at 65 dB, in the presence of 65 dB background noise. A lower ratio than 1 reflects the ability to correctly hear sentences below 65 dB. A ratio higher than 1 reflects the ability to correctly hear sentences presented above 65 dB.
  Manchester and Birmingham are excluded from this analysis due to incorrect set up.
Time Frame: Baseline (unaided) before surgery, 6, 12 and 24 months after surgery
Population: Intention-to-Treat (ITT) population; includes all patient who received the surgical intervention.
  Adaptive Speech in Noise analysis excluded subjects from Birmingham and Manchester clinics due to incorrect set up.
Measure: Mean (Standard Deviation); unit: dB
Arm/Group | Baha Attract System
Number analyzed (Participants) | 36
dB
  SNR 6 months, Baha Attract vs Unaided | -4.30 (5.64)
  SNR 12 months, Baha Attract vs Unaided: number analyzed (Participants) | 35
  SNR 12 months, Baha Attract vs Unaided | 4.79 (6.17)
  SNR 24 months, Baha Attract vs Unaided: number analyzed (Participants) | 31
  SNR 24 months, Baha Attract vs Unaided | -4.47 (6.11)
Statistical Analysis 1: Comparison: Baha Attract System; Speech in Noise, 6 months Baha Attract vs Unaided; Test type: Superiority or Other; p < 0.0001, Fisher's non-parametric permutation test
Statistical Analysis 2: Comparison: Baha Attract System; Speech in Noise, 12 months Baha Attract vs Unaided; Test type: Superiority or Other; p < 0.0001, Fisher's non-parametric permutation test
Statistical Analysis 3: Comparison: Baha Attract System; Speech in Noise, 24 months Baha Attract vs Unaided; Test type: Superiority or Other; p < 0.0001, Fisher's non-parametric permutation test

6. Secondary Outcome: Speech in Quiet, Baha Attract Versus Unaided
Description: The change of hearing performance with the Baha Attract System at 6, 12 and 24 months compared to the pre-operative unaided situation; Speech in quiet at 50, 65 and 80dB.
  Speech in Quiet is a measure of percentage of correct words. A higher score reflects a higher percentage of correct words.
Time Frame: Baseline before surgery, 6, 12 and 24 months after surgery
Population: Intention-to-Treat (ITT) population; includes all patients who received the surgical intervention.
Measure: Mean (Standard Deviation); unit: Change of % correct words at the dB leve
Arm/Group | Baha Attract System
Number analyzed (Participants) | 54
Change of % correct words at the dB leve
  6 months: Speech in quiet at 50dB | 52.1 (29.2)
  6 months: Speech in quiet at 65dB | 43.4 (31.5)
  6 months: Speech in quiet at 80dB | 13.3 (20.6)
  12 months: Speech in quiet at 50dB: number analyzed (Participants) | 51
  12 months: Speech in quiet at 50dB | 50.7 (30.2)
  12 months: Speech in quiet at 65dB: number analyzed (Participants) | 51
  12 months: Speech in quiet at 65dB | 45.5 (31.4)
  12 months: Speech in quiet at 80dB: number analyzed (Participants) | 51
  12 months: Speech in quiet at 80dB | 13.9 (21.2)
  24 months: Speech in quiet at 50dB: number analyzed (Participants) | 46
  24 months: Speech in quiet at 50dB | 40.4 (33.3)
  24 months: Speech in quiet at 65dB: number analyzed (Participants) | 46
  24 months: Speech in quiet at 65dB | 43.3 (29.9)
  24 months: Speech in quiet at 80dB: number analyzed (Participants) | 46
  24 months: Speech in quiet at 80dB | 14.0 (20.7)
Statistical Analysis 1: Comparison: Baha Attract System; 6 months: Speech in quiet at 50dB; Test type: Superiority or Other; p < 0.0001, Fisher's non-parametric permutation test
Statistical Analysis 2: Comparison: Baha Attract System; 6 months: Speech in quiet at 65dB; Test type: Superiority or Other; p < 0.0001, Fisher's non-parametric permutation test
Statistical Analysis 3: Comparison: Baha Attract System; 6 months: Speech in quiet at 80dB; Test type: Superiority or Other; p < 0.0001, Fisher's non-parametric permutation test
Statistical Analysis 4: Comparison: Baha Attract System; 12 months: Speech in quiet at 50dB; Test type: Superiority or Other; p < 0.0001, Fisher's non-parametric permutation test
Statistical Analysis 5: Comparison: Baha Attract System; 12 months: Speech in quiet at 65dB; Test type: Superiority or Other; p < 0.0001, Fisher's non-parametric permutation test
Statistical Analysis 6: Comparison: Baha Attract System; 12 months: Speech in quiet at 80dB; Test type: Superiority or Other; p < 0.0001, Fisher's non-parametric permutation test
Statistical Analysis 7: Comparison: Baha Attract System; 24 months: Speech in quiet at 50dB; Test type: Superiority or Other; p < 0.0001, Fisher's non-parametric permutation test
Statistical Analysis 8: Comparison: Baha Attract System; 24 months: Speech in quiet at 65dB; Test type: Superiority or Other; p < 0.0001, Fisher's non-parametric permutation test
Statistical Analysis 9: Comparison: Baha Attract System; 24 months: Speech in quiet at 80dB; Test type: Superiority or Other; p < 0.0001, Fisher's non-parametric permutation test

7. Secondary Outcome: Hearing Performance: Threshold Audiometry PTA4: Sound Processor on Softband Versus Baha Attract
Description: The change of hearing performance with the Baha Attract System (aided) from the aided hearing performance, sound processor on a softband, before surgery; measured as free-field hearing tests: Threshold audiometry PTA4 (mean of 500, 1000, 2000 and 4000 Hz)
  The units reported for PTA4 are decibels (dB). As such, a lower or more negative score is more desirable and reflects the ability to hear softer sounds.
Time Frame: Baseline before surgery, 6, 12 and 24 months after surgery
Population: Intention-to-Treat (ITT) population; includes all subjects who received the surgical intervention.
Measure: Mean (Standard Deviation); unit: dB
Arm/Group | Baha Attract System
Number analyzed (Participants) | 54
dB
  6 months vs Softband: PTA4 | -0.62 (5.138)
  12 months vs Softband: PTA4: number analyzed (Participants) | 51
  12 months vs Softband: PTA4 | 0.196 (6.719)
  24 months vs Softband: PTA4: number analyzed (Participants) | 46
  24 months vs Softband: PTA4 | -0.136 (6.472)
Statistical Analysis 1: Comparison: Baha Attract System; 6 months with Baha Attract vs Softband: change in PTA4; Test type: Superiority or Other; p = 0.38, Fisher's non-parametric permutation test
Statistical Analysis 2: Comparison: Baha Attract System; 12 months with Baha Attract vs Softband: change in PTA4; Test type: Superiority or Other; p = 0.84, Fisher's non-parametric permutation test
Statistical Analysis 3: Comparison: Baha Attract System; 24 months with Baha Attract vs Softband: change in PTA4; Test type: Superiority or Other; p = 0.89, Fisher's non-parametric permutation test

8. Secondary Outcome: Hearing Performance: Threshold Audiometry Individual Frequencies: Baha Attract Versus Sound Processor on Softband
Description: The change of hearing performance with the Baha Attract System (aided) from the aided hearing performance with Sound processor on a Softband before surgery; measured as free-field hearing tests:
  Threshold audiometry at individual frequencies 250, 500, 1000, 2000, 3000, 4000, 6000 Hz.
  The units reported for threshold audiometry are decibels (dB). As such, a lower or more negative score is more desirable and reflects the ability to hear softer sounds.
Time Frame: Baseline (aided) before surgery, 6 months after surgery
Population: Intention-to-Treat population (ITT); includes all subjects who received the surgical intervention.
Measure: Mean (Standard Deviation); unit: dB
Arm/Group | Baha Attract System
Number analyzed (Participants) | 54
dB
  6 months: Change of Threshold value at 250 Hz | -1.30 (9.77)
  6 months: Change of Threshold value at 500 Hz | -4.17 (7.99)
  6 months: Change of Threshold value at 1000 Hz | -1.11 (6.49)
  6 months: Change of Threshold value at 2000 Hz | -0.463 (7.022)
  6 months: Change of Threshold value at 3000 Hz | 2.69 (9.40)
  6 months: Change of Threshold value at 4000 Hz | 3.24 (9.07)
  6 months: Change of Threshold value at 6000 Hz | 5.56 (9.60)
Statistical Analysis 1: Comparison: Baha Attract System; 250Hz: 6 months with Baha Attract vs Softband; Test type: Superiority or Other; p = 0.34, Fisher's non-parametric permutation test
Statistical Analysis 2: Comparison: Baha Attract System; 500Hz: 6 months with Baha Attract vs Softband; Test type: Superiority or Other; p = 0.0004, Fisher's non-parametric permutation test
Statistical Analysis 3: Comparison: Baha Attract System; 1000Hz: 6 months with Baha Attract vs Softband; Test type: Superiority or Other; p = 0.22, Fisher's non-parametric permutation test
Statistical Analysis 4: Comparison: Baha Attract System; 2000Hz: 6 months with Baha Attract vs Softband; Test type: Superiority or Other; p = 0.64, Fisher's non-parametric permutation test
Statistical Analysis 5: Comparison: Baha Attract System; 3000Hz: 6 months with Baha Attract vs Softband; Test type: Superiority or Other; p = 0.039, Fisher's non-parametric permutation test
Statistical Analysis 6: Comparison: Baha Attract System; 4000Hz: 6 months with Baha Attract vs Softband; Test type: Superiority or Other; p = 0.012, Fisher's non-parametric permutation test
Statistical Analysis 7: Comparison: Baha Attract System; 6000Hz: 6 months with Baha Attract vs Softband; Test type: Superiority or Other; p < 0.0001, Fisher's non-parametric permutation test

9. Secondary Outcome: Hearing Performance: Threshold Audiometry Individual Frequencies: Baha Attract Versus Sound Processor on Softband
Description: The change of hearing performance with the Baha Attract System (aided) from the aided hearing performance with Sound processor on a Softband before surgery; measured as free-field hearing tests:
  Threshold audiometry at individual frequencies: 250, 500, 1000, 2000, 3000, 4000, 6000 Hz.
  The units reported for threshold audiometry are decibels (dB). As such, a lower or more negative score is more desirable and reflects the ability to hear softer sounds.
Time Frame: Baseline (aided) before surgery, 12 months after surgery
Population: Intention-to-Treat population (ITT); includes all subjects who received the surgical intervention.
Measure: Mean (Standard Deviation); unit: dB
Arm/Group | Baha Attract System
Number analyzed (Participants) | 51
dB
  12 months: Change of Threshold value at 250 Hz | -2.55 (11.15)
  12 months: Change of Threshold value at 500 Hz | -2.84 (10.74)
  12 months: Change of Threshold value at 1000 Hz | -0.392 (6.989)
  12 months: Change of Threshold value at 2000 Hz | 0.392 (9.265)
  12 months: Change of Threshold value at 3000 Hz | 4.02 (11.53)
  12 months: Change of Threshold value at 4000 Hz | 3.63 (11.84)
  12 months: Change of Threshold value at 6000 Hz | 5.59 (11.52)
Statistical Analysis 1: Comparison: Baha Attract System; 250Hz: 12 months with Baha Attract vs Softband; Test type: Superiority or Other; p = 0.11, Fisher's non-parametric permutation test
Statistical Analysis 2: Comparison: Baha Attract System; 500Hz: 12 months with Baha Attract vs Softband; Test type: Superiority or Other; p = 0.066, Fisher's non-parametric permutation test
Statistical Analysis 3: Comparison: Baha Attract System; 1000Hz: 12 months with Baha Attract vs Softband; Test type: Superiority or Other; p = 0.71, Fisher's non-parametric permutation test
Statistical Analysis 4: Comparison: Baha Attract System; 2000Hz: 12 months with Baha Attract vs Softband; Test type: Superiority or Other; p = 0.78, Fisher's non-parametric permutation test
Statistical Analysis 5: Comparison: Baha Attract System; 3000Hz: 12 months with Baha Attract vs Softband; Test type: Superiority or Other; p = 0.015, Fisher's non-parametric permutation test
Statistical Analysis 6: Comparison: Baha Attract System; 4000Hz: 12 months with Baha Attract vs Softband; Test type: Superiority or Other; p = 0.035, Fisher's non-parametric permutation test
Statistical Analysis 7: Comparison: Baha Attract System; 6000Hz: 12 months with Baha Attract vs Softband; Test type: Superiority or Other; p = 0.0013, Fisher's non-parametric permutation test

10. Secondary Outcome: Hearing Performance: Threshold Audiometry Individual Frequencies: Baha Attract Versus Sound Processor on Softband
Description: as for outcome 9
Time Frame: Baseline (aided) before surgery, 24 months after surgery
Population: Intention-to-Treat population (ITT); includes all subjects who received the surgical intervention.
Measure: Mean (Standard Deviation); unit: dB
Arm/Group | Baha Attract System
Number analyzed (Participants) | 46
dB
  24 months: Change of Threshold value at 250 Hz: number analyzed (Participants) | 45
  24 months: Change of Threshold value at 250 Hz | -3.67 (8.35)
  24 months: Change of Threshold value at 500 Hz | -1.74 (10.23)
  24 months: Change of Threshold value at 1000 Hz | -1.20 (6.34)
  24 months: Change of Threshold value at 2000 Hz | -0.761 (8.690)
  24 months: Change of Threshold value at 3000 Hz | 2.61 (9.23)
  24 months: Change of Threshold value at 4000 Hz | 3.15 (11.17)
  24 months: Change of Threshold value at 6000 Hz | 5.22 (11.72)
Statistical Analysis 1: Comparison: Baha Attract System; 250Hz: 24 months with Baha Attract vs Softband; Test type: Superiority or Other; p = 0.0051, Fisher's non-parametric permutation test
Statistical Analysis 2: Comparison: Baha Attract System; 500Hz: 24 months with Baha Attract vs Softband; Test type: Superiority or Other; p = 0.26, Fisher's non-parametric permutation test
Statistical Analysis 3: Comparison: Baha Attract System; 1000Hz: 24 months with Baha Attract vs Softband; Test type: Superiority or Other; p = 0.22, Fisher's non-parametric permutation test
Statistical Analysis 4: Comparison: Baha Attract System; 2000Hz: 24 months with Baha Attract vs Softband; Test type: Superiority or Other; p = 0.57, Fisher's non-parametric permutation test
Statistical Analysis 5: Comparison: Baha Attract System; 3000Hz: 24 months with Baha Attract vs Softband; Test type: Superiority or Other; p = 0.064, Fisher's non-parametric permutation test
Statistical Analysis 6: Comparison: Baha Attract System; 4000Hz: 24 months with Baha Attract vs Softband; Test type: Superiority or Other; p = 0.064, Fisher's non-parametric permutation test
Statistical Analysis 7: Comparison: Baha Attract System; 6000Hz: 24 months with Baha Attract vs Softband; Test type: Superiority or Other; p = 0.0051, Fisher's non-parametric permutation test

11. Secondary Outcome: Adaptive Speech Recognition in Noise Ratio: Baha Attract Versus Sound Processor on Softband
Description: The change of hearing performance with the Baha Attract System compared to the pre-operative aided situation with Sound Processor on a softband; Adaptive Speech recognition in Noise measured as signal to noise ratio.
  A ratio of 1 reflects the ability to correctly hear sentences at 65 dB, in the presence of 65 dB background noise. A lower ratio than 1 reflects the ability to correctly hear sentences below 65 dB. A ratio higher than 1 reflects the ability to correctly hear sentences presented above 65 dB.
Time Frame: Baseline (aided) before surgery, 6, 12 and 24 months after surgery
Population: Intention-to-Treat (ITT) population; includes all patient who received the surgical intervention.
  Speech in Noise analysis excludes patients from Birmingham and Manchester due to incorrect set up.
Measure: Mean (Standard Deviation); unit: change in SNR dB
Arm/Group | Baha Attract System
Number analyzed (Participants) | 38
change in SNR dB
  6 months: Speech in Noise | -0.508 (4.173)
  12 months: Speech in Noise: number analyzed (Participants) | 37
  12 months: Speech in Noise | -1.05 (4.75)
  24 months: Speech in Noise: number analyzed (Participants) | 33
  24 months: Speech in Noise | -0.739 (4.106)
Statistical Analysis 1: Comparison: Baha Attract System; 6 months: Speech in Noise with Baha Attract vs Softband; Test type: Superiority or Other; p = 0.46, Fisher's non-parametric permutation test
Statistical Analysis 2: Comparison: Baha Attract System; 12 months: Speech in Noise with Baha Attract vs Softband; Test type: Superiority or Other; p = 0.19, Fisher's non-parametric permutation test
Statistical Analysis 3: Comparison: Baha Attract System; 24 months: Speech in Noise with Baha Attract vs Softband; Test type: Superiority or Other; p = 0.31, Fisher's non-parametric permutation test

12. Secondary Outcome: Speech in Quiet: Baha Attract Versus Sound Processor on Softband
Description: The change of hearing performance with the Baha Attract System at 6 months compared to the pre-operative aided situation with the Sound Processor on a softband; Speech in quiet at 50, 65 and 80dB.
  Speech in Quiet is a measure of percentage of correct words. A higher score reflects a higher percentage of correct words.
Time Frame: Baseline (aided) before surgery, 6, 12 and 24 months after surgery
Population: Intention-to-Treat (ITT) population; includes all patients who received the surgical intervention.
Measure: Mean (Standard Deviation); unit: Change of % correct words at the dB leve
Arm/Group | Baha Attract System
Number analyzed (Participants) | 54
Change of % correct words at the dB leve
  6 months: Speech in quiet at 50dB | 2.74 (29.94)
  6 months: Speech in quiet at 65dB | -2.11 (10.62)
  6 months: Speech in quiet at 80dB | -0.33 (5.00)
  12 months: Speech in quiet at 50dB: number analyzed (Participants) | 51
  12 months: Speech in quiet at 50dB | 0.373 (27.201)
  12 months: Speech in quiet at 65dB: number analyzed (Participants) | 51
  12 months: Speech in quiet at 65dB | -2.69 (11.16)
  12 months: Speech in quiet at 80dB: number analyzed (Participants) | 51
  12 months: Speech in quiet at 80dB | -0.961 (8.457)
  24 months: Speech in quiet at 50dB: number analyzed (Participants) | 46
  24 months: Speech in quiet at 50dB | -11.6 (32.6)
  24 months: Speech in quiet at 65dB: number analyzed (Participants) | 46
  24 months: Speech in quiet at 65dB | -5.67 (16.48)
  24 months: Speech in quiet at 80dB: number analyzed (Participants) | 46
  24 months: Speech in quiet at 80dB | -0.696 (8.178)
Statistical Analysis 1: Comparison: Baha Attract System; 6 months Speech in Quiet at 50dB; Test type: Superiority or Other; p = 0.43, Fisher's non-parametric permutation test
Statistical Analysis 2: Comparison: Baha Attract System; 6 months Speech in Quiet at 65dB; Test type: Superiority or Other; p = 0.16, Fisher's non-parametric permutation test
Statistical Analysis 3: Comparison: Baha Attract System; 6 months Speech in Quiet at 80dB; Test type: Superiority or Other; p = 0.65, Fisher's non-parametric permutation test
Statistical Analysis 4: Comparison: Baha Attract System; 12 months Speech in Quiet at 50dB; Test type: Superiority or Other; p = 0.93, Fisher's non-parametric permutation test
Statistical Analysis 5: Comparison: Baha Attract System; 12 months Speech in Quiet at 65dB; Test type: Superiority or Other; p = 0.094, Fisher's non-parametric permutation test
Statistical Analysis 6: Comparison: Baha Attract System; 12 months Speech in Quiet at 80dB; Test type: Superiority or Other; p = 0.44, Fisher's non-parametric permutation test
Statistical Analysis 7: Comparison: Baha Attract System; 24 months Speech in Quiet at 50dB; Test type: Superiority or Other; p = 0.021, Fisher's non-parametric permutation test
Statistical Analysis 8: Comparison: Baha Attract System; 24 months Speech in Quiet at 65dB; Test type: Superiority or Other; p = 0.024, Fisher's non-parametric permutation test
Statistical Analysis 9: Comparison: Baha Attract System; 24 months Speech in Quiet at 80dB; Test type: Superiority or Other; p = 0.59, Fisher's non-parametric permutation test

13. Secondary Outcome: Health Utility Index (HUI)
Description: Change of health status and health related quality of life using the generic quality of life scale Health Utilities Index (HUI3) when wearing Baha Attract System compared to the pre-operative unaided situation. A health utility value of 1.00 indicates perfect health while a score of 0.00 indicates death. The change from unaided to aided hearing is presented. A positive value indicates an improved quality of life, a negative value indicates impaired quality of life.
  HUI score of 1 (maximum) describes a state of perfect health. HUI score of 0 describes a state of dead. A negative score of Comprehensive Health State describes a state worse than dead.
Time Frame: Baseline (unaided) before surgery, 6 and 24 months after surgery
Population: Intention-to-Treat (ITT) population; includes all patients who received the surgical intervention.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Baha Attract System
Number analyzed (Participants) | 53
units on a scale
  6 months: Comprehensive health state: number analyzed (Participants) | 47
  6 months: Comprehensive health state | 0.063 (0.249)
  6 months: Vision | -0.003 (0.033)
  6 months: Hearing: number analyzed (Participants) | 49
  6 months: Hearing | 0.111 (0.321)
  6 months: Speech: number analyzed (Participants) | 52
  6 months: Speech | 0.045 (0.153)
  6 months: Ambulation | -0.016 (0.067)
  6 months: Dexterity | -0.021 (0.108)
  6 months: Emotion | 0.017 (0.152)
  6 months: Cognition: number analyzed (Participants) | 52
  6 months: Cognition | 0.005 (0.158)
  6 months: Pain | 0.020 (0.123)
  24 months: Comprehensive health state: number analyzed (Participants) | 37
  24 months: Comprehensive health state | 0.069 (0.240)
  24 months: Vision: number analyzed (Participants) | 46
  24 months: Vision | 0.002 (0.015)
  24 months: Hearing: number analyzed (Participants) | 39
  24 months: Hearing | 0.119 (0.358)
  24 months: Speech: number analyzed (Participants) | 44
  24 months: Speech | 0.051 (0.135)
  24 months: Ambulation: number analyzed (Participants) | 46
  24 months: Ambulation | -0.015 (0.076)
  24 months: Dexterity: number analyzed (Participants) | 44
  24 months: Dexterity | -0.025 (0.151)
  24 months: Emotion: number analyzed (Participants) | 44
  24 months: Emotion | 0.014 (0.089)
  24 months: Cognition: number analyzed (Participants) | 45
  24 months: Cognition | 0.003 (0.134)
  24 months: Pain: number analyzed (Participants) | 45
  24 months: Pain | 0.040 (0.117)
Statistical Analysis 1: Comparison: Baha Attract System; 6 months change in Comprehensive health state; Test type: Superiority or Other; p = 0.088, Fisher's non-parametric permutation test
Statistical Analysis 2: Comparison: Baha Attract System; 6 months change in Vision; Test type: Superiority or Other; p = 0.88, Fisher's non-parametric permutation test
Statistical Analysis 3: Comparison: Baha Attract System; 6 months change in Hearing; Test type: Superiority or Other; p = 0.020, Fisher's non-parametric permutation test
Statistical Analysis 4: Comparison: Baha Attract System; 6 months change in Speech; Test type: Superiority or Other; p = 0.039, Fisher's non-parametric permutation test
Statistical Analysis 5: Comparison: Baha Attract System; 6 months change in Ambulation; Test type: Superiority or Other; p = 0.25, Fisher's non-parametric permutation test
Statistical Analysis 6: Comparison: Baha Attract System; 6 months change in Dexterity; Test type: Superiority or Other; p = 0.38, Fisher's non-parametric permutation test
Statistical Analysis 7: Comparison: Baha Attract System; 6 months change in Emotion; Test type: Superiority or Other; p = 0.43, Fisher's non-parametric permutation test
Statistical Analysis 8: Comparison: Baha Attract System; 6 months change in Cognition; Test type: Superiority or Other; p = 0.85, Fisher's non-parametric permutation test
Statistical Analysis 9: Comparison: Baha Attract System; 6 months change in Pain; Test type: Superiority or Other; p = 0.25, Fisher's non-parametric permutation test
Statistical Analysis 10: Comparison: Baha Attract System; 24 months change in Comprehensive health state; Test type: Superiority or Other; p = 0.088, Fisher's non-parametric permutation test
Statistical Analysis 11: Comparison: Baha Attract System; 24 months change in Vision; Test type: Superiority or Other; p = 0.63, Fisher's non-parametric permutation test
Statistical Analysis 12: Comparison: Baha Attract System; 24 months change in Hearing; Test type: Superiority or Other; p = 0.045, Fisher's non-parametric permutation test
Statistical Analysis 13: Comparison: Baha Attract System; 24 months change in Speech; Test type: Superiority or Other; p = 0.016, Fisher's non-parametric permutation test
Statistical Analysis 14: Comparison: Baha Attract System; 24 months change in Ambulation; Test type: Superiority or Other; p = 0.25, Fisher's non-parametric permutation test
Statistical Analysis 15: Comparison: Baha Attract System; 24 months change in Dexterity; Test type: Superiority or Other; p = 0.50, Wilcoxan Signed Rank Test; Fisher's non-parametric permutation test failed to approximate p value so Wilcoxan Signed Rank Test instead
Statistical Analysis 16: Comparison: Baha Attract System; 24 months change in Emotion; Test type: Superiority or Other; p = 0.29, Fisher's non-parametric permutation test
Statistical Analysis 17: Comparison: Baha Attract System; 24 months change in Cognition; Test type: Superiority or Other; p = 0.92, Fisher's non-parametric permutation test
Statistical Analysis 18: Comparison: Baha Attract System; 24 months change in Pain; Test type: Superiority or Other; p = 0.020, Fisher's non-parametric permutation test

14. Secondary Outcome: Abbreviated Profile of Hearing Aid Benefit (APHAB)
Description: Measuring change of Ease of communication, Reverberation, Background noise, Aversiveness and a Global score with the Baha Attract System from the pre-operative unaided situation. The absolute APHAB scale is between 0 and 100%, where 0% indicates no problems and 100% indicates always problem. The change from unaided to aided hearing is presented. A positive value indicates an improvement, a negative value an impairment.
Time Frame: Baseline before surgery, 6 and 24 months after surgery
Population: Intention-to-Treat (ITT) population; includes all patients who received the surgical intervention.
Measure: Mean (Standard Deviation); unit: units on scale
Arm/Group | Baha Attract System
Number analyzed (Participants) | 53
units on scale
  6 months: Ease of communication | 20.4 (24.9)
  6 months: Background noise | 26.3 (20.6)
  6 months: Reverberation | 22.0 (19.0)
  6 months: Aversiveness | 1.32 (23.45)
  6 months: Global | 22.9 (18.1)
  24 months: Ease of communication: number analyzed (Participants) | 45
  24 months: Ease of communication | 18.7 (26.3)
  24 months: Background noise: number analyzed (Participants) | 45
  24 months: Background noise | 23.7 (20.4)
  24 months: Reverberation: number analyzed (Participants) | 45
  24 months: Reverberation | 20.8 (19.9)
  24 months: Aversiveness: number analyzed (Participants) | 45
  24 months: Aversiveness | -0.596 (19.646)
  24 months: Global: number analyzed (Participants) | 45
  24 months: Global | 21.1 (18.9)
Statistical Analysis 1: Comparison: Baha Attract System; 6 months: Ease of communication; Test type: Superiority or Other; p < 0.0001, Fisher's non-parametric permutation test
Statistical Analysis 2: Comparison: Baha Attract System; 6 months: Background noise; Test type: Superiority or Other; p < 0.0001, Fisher's non-parametric permutation test
Statistical Analysis 3: Comparison: Baha Attract System; 6 months: Reverberation; Test type: Superiority or Other; p < 0.0001, Fisher's non-parametric permutation test
Statistical Analysis 4: Comparison: Baha Attract System; 6 months: Aversiveness; Test type: Superiority or Other; p = 0.69, Fisher's non-parametric permutation test
Statistical Analysis 5: Comparison: Baha Attract System; 6 months: Global; Test type: Superiority or Other; p < 0.0001, Fisher's non-parametric permutation test
Statistical Analysis 6: Comparison: Baha Attract System; 24 months: Ease of communication; Test type: Superiority or Other; p < 0.001, Fisher's non-parametric permutation test
Statistical Analysis 7: Comparison: Baha Attract System; 24 months: Background noise; Test type: Superiority or Other; p < 0.001, Fisher's non-parametric permutation test
Statistical Analysis 8: Comparison: Baha Attract System; 24 months: Reverberation; Test type: Superiority or Other; p < 0.001, Fisher's non-parametric permutation test
Statistical Analysis 9: Comparison: Baha Attract System; 24 months: Aversiveness; Test type: Superiority or Other; p = 0.84, Fisher's non-parametric permutation test
Statistical Analysis 10: Comparison: Baha Attract System; 24 months: Global; Test type: Superiority or Other; p < 0.001, Fisher's non-parametric permutation test; Fisher's non-parametric permutation test

15. Secondary Outcome: Speech, Spatial and Qualities of Hearing Scale (SSQ)
Description: Measuring change of speech, spatial and hearing experiences with the Baha Attract System from the pre-operative unaided situation. A scale from 0 to 10, where 0 represents "can not hear at all", and 10 "hear perfectly". The change from unaided to aided hearing is presented. A positive value indicates improved hearing, a negative value indicates impaired hearing.
Time Frame: Baseline before surgery, 6 and 24 months after surgery
Population: Intention-to-Treat (ITT) population; includes all patient who received the surgical intervention.
Measure: Mean (Standard Deviation); unit: units on scale
Arm/Group | Baha Attract System
Number analyzed (Participants) | 53
units on scale
  Speech: Change from pre-op to 6 months | 2.49 (1.67)
  Spatial: Change from pre-op to 6 months | 1.87 (1.90)
  Qualities: Change from pre-op to 6 months | 1.68 (1.36)
  Speech: Change from pre-op to 24 months: number analyzed (Participants) | 46
  Speech: Change from pre-op to 24 months | 2.07 (1.57)
  Spatial: Change from pre-op to 24 months: number analyzed (Participants) | 46
  Spatial: Change from pre-op to 24 months | 1.36 (1.74)
  Qualities: Change from pre-op to 24 months: number analyzed (Participants) | 46
  Qualities: Change from pre-op to 24 months | 1.30 (1.39)
Statistical Analysis 1: Comparison: Baha Attract System; Speech: Change from pre-op to 6 months; Test type: Superiority or Other; p < 0.0001, Fisher's non-parametric permutation test
Statistical Analysis 2: Comparison: Baha Attract System; Spatial: Change from pre-op to 6 months; Test type: Superiority or Other; p < 0.0001, Fisher's non-parametric permutation test
Statistical Analysis 3: Comparison: Baha Attract System; Qualities: Change from pre-op to 6 months; Test type: Superiority or Other; p < 0.0001, Fisher's non-parametric permutation test
Statistical Analysis 4: Comparison: Baha Attract System; Speech: Change from pre-op to 24 months; Test type: Superiority or Other; p < 0.0001, Fisher's non-parametric permutation test
Statistical Analysis 5: Comparison: Baha Attract System; Spatial: Change from pre-op to 24 months; Test type: Superiority or Other; p < 0.0001, Fisher's non-parametric permutation test
Statistical Analysis 6: Comparison: Baha Attract System; Qualities: Change from pre-op to 24 months; Test type: Superiority or Other; p < 0.0001, Fisher's non-parametric permutation test

16. Secondary Outcome: Time to Perform Surgery
Description: Time of first incision to time of last suture
Time Frame: Visit 2 (Surgery)
Population: Intention-to-Treat (ITT) population; includes all patients who received the surgical intervention.
Measure: Mean (Standard Deviation); unit: Minutes
Arm/Group | Baha Attract System
Number analyzed (Participants) | 54
Minutes | 38.7 (10.7)

17. Secondary Outcome: Tissue Reduction Performed During Surgery
Description: Surgical thinning of the soft tissue flap was advocated when the soft tissue thickness exceeded 6 mm
Time Frame: Visit 2 (surgery)
Population: Intention-to-Treat (ITT) population; all patients who received surgical intervention.
Measure: Number; unit: participants
Arm/Group | Baha Attract System
Number analyzed (Participants) | 54
participants
  Tissue thinning | 12
  No tissue thinning | 42

18. Secondary Outcome: Implant Stability
Description: Implant Stability Quotient - ISQ, a scale from 1 to 100, where 100 represent the highest stability
Time Frame: Visit 2 (surgery)
Population: Intention-to-treat (ITT) population; includes all patients who received surgical intervention.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Baha Attract System
Number analyzed (Participants) | 54
units on a scale | 77.3 (9.0)

19. Secondary Outcome: Magnetic Force
Description: To investigate if the magnetic force required for sound processor magnet retention will change over time
Time Frame: 4, 6, 12 weeks, 6, 12 and 24 months
Population: Intention-to-Treat (ITT) population; includes all patients who received surgical intervention.
Measure: Mean (Standard Deviation); unit: Newton
Arm/Group | Baha Attract System
Number analyzed (Participants) | 54
Newton
  4 weeks | 1.01 (0.40)
  6 weeks: number analyzed (Participants) | 53
  6 weeks | 1.07 (0.33)
  12 weeks: number analyzed (Participants) | 53
  12 weeks | 1.15 (0.41)
  6 months: number analyzed (Participants) | 53
  6 months | 1.16 (0.42)
  12 months: number analyzed (Participants) | 52
  12 months | 1.15 (0.38)
  24 months: number analyzed (Participants) | 47
  24 months | 1.09 (0.41)

20. Secondary Outcome: Sound Processor Magnet Choice
Description: To investigate how sound processor magnet choice will change over time. Six different magnetic strength could be chosen; SPM 1 had the lowest strength and SPM 6 the the highest.
Time Frame: 4, 6, 12 weeks, 6, 12 and 24 months
Population: Intention-to-Treat (ITT) population; includes all patients who received surgical intervention at week 4. At week 6, 12 and month 6, 12 and 24 one patient had left the study.
Measure: Count of Participants; unit: Participants
Arm/Group | Baha Attract System
Number analyzed (Participants) | 54
Participants
  Week 4: SPM 6 | 19
  Week 4: SPM 5 | 19
  Week 4: SPM 4 | 9
  Week 4: SPM 3 | 6
  Week 4: SPM 2 | 1
  Week 4: SPM 1 | 0
  Week 6: number analyzed (Participants) | 53
  Week 6: SPM 6 | 11
  Week 6: SPM 5 | 10
  Week 6: SPM 4 | 16
  Week 6: SPM 3 | 13
  Week 6: SPM 2 | 2
  Week 6: SPM 1 | 1
  Week 12: number analyzed (Participants) | 53
  Week 12: SPM 6 | 6
  Week 12: SPM 5 | 12
  Week 12: SPM 4 | 11
  Week 12: SPM 3 | 15
  Week 12: SPM 2 | 9
  Week 12: SPM 1 | 0
  Month 6: number analyzed (Participants) | 53
  Month 6: SPM 6 | 5
  Month 6: SPM 5 | 9
  Month 6: SPM 4 | 12
  Month 6: SPM 3 | 18
  Month 6: SPM 2 | 9
  Month 6: SPM 1 | 0
  Month 12: number analyzed (Participants) | 52
  Month 12: SPM 6 | 6
  Month 12: SPM 5 | 11
  Month 12: SPM 4 | 12
  Month 12: SPM 3 | 14
  Month 12: SPM 2 | 8
  Month 12: SPM 1 | 1
  Month 24: number analyzed (Participants) | 46
  Month 24: SPM 6 | 5
  Month 24: SPM 5 | 8
  Month 24: SPM 4 | 5
  Month 24: SPM 3 | 17
  Month 24: SPM 2 | 9
  Month 24: SPM 1 | 2

21. Secondary Outcome: Pain & Discomfort
Description: Degree of pain and discomfort.
Time Frame: Week 6, Week 12, Month 6, Month 12, Month 24
Population: Safety population; includes all patients who received the surgical intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | Baha Attract System
Number analyzed (Participants) | 54
Participants
  Week 6: number analyzed (Participants) | 53
  Week 6: No Discomfort or Pain | 21
  Week 6: Slight Discomfort or Pain | 15
  Week 6: Discomfort or Pain | 15
  Week 6: Excessive Discomfort or Pain | 2
  Week 12: number analyzed (Participants) | 53
  Week 12: No Discomfort or Pain | 24
  Week 12: Slight Discomfort or Pain | 16
  Week 12: Discomfort or Pain | 11
  Week 12: Excessive Discomfort or Pain | 2
  Month 6: number analyzed (Participants) | 53
  Month 6: No Discomfort or Pain | 33
  Month 6: Slight Discomfort or Pain | 15
  Month 6: Discomfort or Pain | 5
  Month 6: Excessive Discomfort or Pain | 0
  Month 12: number analyzed (Participants) | 52
  Month 12: No Discomfort or Pain | 37
  Month 12: Slight Discomfort or Pain | 11
  Month 12: Discomfort or Pain | 4
  Month 12: Excessive Discomfort or Pain | 0
  Month 24: number analyzed (Participants) | 47
  Month 24: No Discomfort or Pain | 40
  Month 24: Slight Discomfort or Pain | 4
  Month 24: Discomfort or Pain | 3
  Month 24: Excessive Discomfort or Pain | 0

22. Secondary Outcome: Numbness When Tested With a Pin
Description: Degree of numbness when tested with a pin
Time Frame: Day 10, Week 4, Week 6, Week 12, Month 6, Month 12, Month 24
Population: Safety population; includes all patients who received the surgical intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | Baha Attract System
Number analyzed (Participants) | 54
Participants
  Day 10: Numbness tested with a Pin: No Numbness | 12
  Day 10: Numbness tested with a Pin: Numbness within 2cm of Implant | 9
  Day 10: Numbness tested with a Pin: Numbness within & beyond 2cm from Implant | 33
  Week 4: Numbness tested with a pin: No Numbness | 15
  Week 4: Numbness tested with a pin: Numbness within 2cm of Implant | 7
  Week 4: Numbness tested with a pin: Numbness within & beyond 2cm from Implant | 32
  Week 6: Numbness tested with a pin: number analyzed (Participants) | 53
  Week 6: Numbness tested with a pin: No Numbness | 21
  Week 6: Numbness tested with a pin: Numbness within 2cm of Implant | 3
  Week 6: Numbness tested with a pin: Numbness within & beyond 2cm from Implant | 29
  Week 12: Numbness tested with a pin: number analyzed (Participants) | 53
  Week 12: Numbness tested with a pin: No Numbness | 33
  Week 12: Numbness tested with a pin: Numbness within 2cm of Implant | 5
  Week 12: Numbness tested with a pin: Numbness within & beyond 2cm from Implant | 15
  Month 6: Numbness tested with a Pin: number analyzed (Participants) | 52
  Month 6: Numbness tested with a Pin: No Numbness | 42
  Month 6: Numbness tested with a Pin: Numbness within 2cm of Implant | 3
  Month 6: Numbness tested with a Pin: Numbness within & beyond 2cm from Implant | 7
  Month 12: Numbness tested with a Pin: number analyzed (Participants) | 52
  Month 12: Numbness tested with a Pin: No Numbness | 45
  Month 12: Numbness tested with a Pin: Numbness within 2cm of Implant | 3
  Month 12: Numbness tested with a Pin: Numbness within & beyond 2cm from Implant | 4
  Month 24: Numbness tested with a Pin: number analyzed (Participants) | 46
  Month 24: Numbness tested with a Pin: No Numbness | 45
  Month 24: Numbness tested with a Pin: Numbness within 2cm of Implant | 0
  Month 24: Numbness tested with a Pin: Numbness within & beyond 2cm from Implant | 1

23. Secondary Outcome: Numbness When Tested With a Cotton Swab
Description: Degree of numbness when tested with a Cotton Swab
Time Frame: Day 10, Week 4, Week 6, Week 12, Month 6, Month 12, Month 24
Population: Safety population; includes all patients who received the surgical intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | Baha Attract System
Number analyzed (Participants) | 54
Participants
  Day 10: Numbness tested with a Cotton Swab: No Numbness | 13
  Day 10: Numbness tested with a Cotton Swab: Numbness within 2 cm from implant | 9
  Day 10: Numbness tested with a Cotton Swab: Numbness within & beyond 2cm from Implant | 32
  Week 4: Numbness tested with a Cotton Swab: No Numbness | 18
  Week 4: Numbness tested with a Cotton Swab: Numbness within 2 cm from implant | 6
  Week 4: Numbness tested with a Cotton Swab: Numbness within & beyond 2cm from Implant | 30
  Week 6: Numbness tested with a Cotton Swab: number analyzed (Participants) | 53
  Week 6: Numbness tested with a Cotton Swab: No Numbness | 23
  Week 6: Numbness tested with a Cotton Swab: Numbness within 2 cm from implant | 2
  Week 6: Numbness tested with a Cotton Swab: Numbness within & beyond 2cm from Implant | 28
  Week 12: Numbness tested with a Cotton Swab: number analyzed (Participants) | 53
  Week 12: Numbness tested with a Cotton Swab: No Numbness | 31
  Week 12: Numbness tested with a Cotton Swab: Numbness within 2 cm from implant | 6
  Week 12: Numbness tested with a Cotton Swab: Numbness within & beyond 2cm from Implant | 16
  Month 6: Numbness tested with a Cotton Swab: number analyzed (Participants) | 52
  Month 6: Numbness tested with a Cotton Swab: No Numbness | 43
  Month 6: Numbness tested with a Cotton Swab: Numbness within 2 cm from implant | 2
  Month 6: Numbness tested with a Cotton Swab: Numbness within & beyond 2cm from Implant | 7
  Month 12: Numbness tested with a Cotton Swab: number analyzed (Participants) | 52
  Month 12: Numbness tested with a Cotton Swab: No Numbness | 44
  Month 12: Numbness tested with a Cotton Swab: Numbness within 2 cm from implant | 3
  Month 12: Numbness tested with a Cotton Swab: Numbness within & beyond 2cm from Implant | 5
  Month 24: Numbness tested with a Cotton Swab: number analyzed (Participants) | 46
  Month 24: Numbness tested with a Cotton Swab: No Numbness | 42
  Month 24: Numbness tested with a Cotton Swab: Numbness within 2 cm from implant | 3
  Month 24: Numbness tested with a Cotton Swab: Numbness within & beyond 2cm from Implant | 1

ADVERSE EVENTS:
Time Frame: 24 months
Description: The AEs were encoded according to the CTCAE dictionary and only to the SOC term.
Arm/Group | Baha Attract System
All-Cause Mortality (participants affected / at risk) | 1/54
Serious Adverse Events (participants affected / at risk) | 13/54
Other Adverse Events (participants affected / at risk) | 29/54
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Baha Attract System (N=54)
Infection (Infections and infestations) | 1 (1) — Adverse Event Term is the Reported term
Increase in instability of knee prosthesis (General disorders) | 1 (1) — Adverse Event Term is the Reported term
Pancreatitis (Gastrointestinal disorders) | 1 (1) — Adverse Event Term is the Reported term
Embolisation of the Splenic Artery from pancreatitis (Blood and lymphatic system disorders) | 1 (1) — Adverse Event Term is the Reported term
Increase of Meniere Attacks (Ear and labyrinth disorders) | 1 (1) — Adverse Event Term is the Reported term
Progression of Hearing Loss (Ear and labyrinth disorders) | 1 (1) — Adverse Event Term is the Reported term
Decompensated Alcoholic Liver Disease (Hepatobiliary disorders) | 1 (1) — Adverse Event Term is the Reported term
Broken Ankle (Injury, poisoning and procedural complications) | 1 (1) — Adverse Event Term is the Reported term
Cholesteatoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) — Adverse Event Term is the Reported term
Pain/Discomfort (Injury, poisoning and procedural complications) | 1 (1) — Adverse Event Term is the Reported term
Surgery for Baha Attract on other ear (Surgical and medical procedures) | 1 (1) — Adverse Event Term is the Reported term
Increase in Occlusive Arterial Disease (Vascular disorders) | 1 (1) — Adverse Event Term is the Reported term
Dequervian (Musculoskeletal and connective tissue disorders) | 1 (1) — Adverse Event Term is the Reported term
Patient was addmitted to the hospital due to childbirth (Pregnancy, puerperium and perinatal conditions) | 1 (1) — Adverse Event Term is the Reported term
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Baha Attract System (N=54)
Ear and Labyrinth Disorders (Ear and labyrinth disorders) | 6 (9)
Gastrointestinal Disorders (Gastrointestinal disorders) | 4 (5)
General Disorders and Administration Site Conditions (General disorders) | 10 (10)
Infections and Infestation (Infections and infestations) | 14 (21)
Injury, Poisoning and Procedural Complications (Infections and infestations) | 5 (5)
Musculoskeletal and Connective Tissue Disorders (Musculoskeletal and connective tissue disorders) | 4 (4)
Nervous System Disorders (Nervous system disorders) | 5 (5)
Respiratory, Thoracic and Mediastinal Disorders (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Skin and Subcutaneous Tissue Disorders (Skin and subcutaneous tissue disorders) | 7 (7)
Vascular Disorders (Vascular disorders) | 3 (3)
Predefined event: Pressure related Skin Complications (Skin and subcutaneous tissue disorders) | 6 (6)
Predefined event: Pain/Discomfort (Skin and subcutaneous tissue disorders) | 24 (37)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2013-11-22): https://cdn.clinicaltrials.gov/large-docs/85/NCT02022085/Prot_000.pdf
  • Statistical Analysis Plan (2016-02-26): https://cdn.clinicaltrials.gov/large-docs/85/NCT02022085/SAP_001.pdf